CLINICAL TRIAL: NCT06657378
Title: A Multicenter, Postmarketing Observational (Noninterventional) Study to Evaluate the Safety of Fycompa for Injection in Patients With Partial-Onset Seizures (Including Secondarily Generalized Seizures) (Age 4 Years or Older) or Primary Generalized Tonic- Clonic Seizures (Age 12 Years or Older)
Brief Title: A Study to Evaluate the Safety of Fycompa Injection in Participants With Partial-Onset Seizures or Primary Generalized Tonic- Clonic Seizures
Status: Recruiting | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2007-M081-517
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Partial-Onset Seizures; Primary Generalized Tonic-clonic Seizures
Keywords: Seizures; Secondarily Generalized Seizures; Fycompa
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fycompa
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The purpose of this study is to determine the safety of Fycompa for injection after administration in participants with epilepsy (partial-onset seizures [including secondarily generalized seizures]) (age 4 years or older) or primary generalized tonic-clonic seizures (age 12 years or older).

ELIGIBILITY:
Inclusion Criteria:

* Participants with epilepsy who received the Fycompa for injection for the first time will be included.

Exclusion Criteria:

* The exclusion criteria will not be specified in particular because this survey will be conducted in daily clinical practice.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with epilepsy who received the Fycompa for injection for the first time will be included.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Drug Reactions (ADRs) and Adverse Events (AEs) | Up to 4 weeks
Number of Participants With ADRs Based on Participant Characteristic | Up to 4 weeks
Plasma Concentration of Fycompa in Children Aged Greater Than or Equal to (>=) 4 Years and Less than (<) 12 Years | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 1, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.